CLINICAL TRIAL: NCT00157508
Title: A Pilot, Randomised, Double-blind, Cross-over Study to Assess the Renal and Systemic Effects of NCX4016 in Patients With Type 2 Diabetes and Early Nephropathy
Brief Title: Renal and Systemic Effects of NCX4016 in Patients With Type 2 Diabetes and Early Nephropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NCX4016-X-204
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2005-09

CONDITIONS: Type 2 Diabetes; Early Nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Diseases | interventions — nitroaspirin

INTERVENTIONS:
Drug: nitroaspirin

SUMMARY:
Aspirin is commonly used for treatment of painful and inflammatory diseases and in the prevention of the cardiovascular disease. A major drawback of aspirin treatment is the well recognized gastrointestinal toxicity. Recent research indicate that coupling a nitric oxide (NO)derivate to the aspirin moiety retains its therapeutic effects while avoiding its undesirable gastrointestinal side effects. NO has cytoprotective effects, such as blood flow modulation, mucus release and repair of mucosal injury. NCX4016, a NO-releasing derivative of acetylsalicilic acid, has been shown to retain the analgesic, anti-inflammatory and antithrombotic activity of aspirin, but with less gastrointestinal toxicity. In addition, preliminary data suggested that NCX4016 may restore insulin sensitivity in eNOS deficient mice.

This study was aimed to evaluate the activity of NCX4016, compared to aspirin, on albuminuria, insulin sensitivity and cardiac and renal hemodynamic in patients with type 2 diabetes mellitus. The patients after one month of placebo treatment, entered two 1-month treatments periods, with equivalent doses (800 mg of NCX4016, 325 mg of aspirin) of NCX4016 or aspirin.

DETAILED DESCRIPTION:
Nitric oxide-releasing, non-steroidal anti-inflammatory drugs (NO-NSAIDs) are new chemical entities obtained by adding a nitric oxide-releasing moiety to the parent NSAID via a short-chain ester linkage. NCX4016 (Nitro-aspirin), a acetoxy-benzoate 2-(2-nitroxymethyl)-phenyl ester of acetylsalicylic acid, is one of these novel compounds developed with the dual aim to expand the pharmacological properties of the parent drug and to spare some of its side effects, in particular on the gastrointestinal mucosa. Decreased NO synthesis may contribute to some of the abnormalities associated with diabetes such as decreased insulin activity, impaired endothelium-dependent/insulin-induced vasodilatation, increased sympathetic vasoconstrictor outflow and increased platelet activation, that may result in increased vascular resistance and arterial hypertension and, in the long term, to an increased risk of micro- and macrovascular complications.

Low-dose aspirin represents the antiplatelet drug of choice for prevention of vascular complications in diabetes. Preclinical data on NCX4016 support the possibility that Nitro-aspirin may shear with aspirin the antithrombotic activity and may offer the additional benefits related to increased NO bioavailability. Actually NCX4016 inhibits cyclooxygenase (COX) activity in platelets both in vitro and ex vivo and, similar to aspirin, prevents the release of thromboxane (TX) A2 and arachidonic acid-induced platelet aggregation. Moreover Nitro-aspirin inhibits aspirin-insensitive platelet aggregation and adhesion, possibly by inhibiting the expression of platelet adhesion molecules by a specific COX-independent mechanism, probably NO-mediated, that is not show by the parent compound. Therefore Nitro-aspirin can exceed the cardioprotective action of the parent compound, by adding the aspirin-like moiety and the NO-releasing moiety, which both contribute to its benefits effects, such as multiple anti-thrombotic and, possibly, anti-atherosclerotic activities, restoration of insulin-related metabolic and vascular effect and finally blood pressure reduction. Moreover, experimental and clinical data suggest that Nitro-aspirin will offer significant safety advantages by its NO moiety that may limit aspirin gastrotoxicity by preventing the vasocontriction of the mucosal microvasculature.

In the present randomised, double-blind, cross-over study, we evaluated the efficacy and safety profile of Nitro-aspirin (800 mg bid), and of an equiactive dose of aspirin (325 mg od), as compared to placebo, in thirteen patients with type 2 diabetes and micro or macro-albuminuria (overnight albumin excretion rate > 20 µg/min for at least 6 months), without overt renal insufficiency (serum creatinine concentration < 2 mg/dl) and no specific controindication to aspirin therapy. Eligible patients who provided written informed consent, withdrew any previous treatment with NSAIDs or aspirin and, after a 4-week placebo run-in period, entered two consecutive 4-week treatment periods with Nitro-aspirin plus aspirin placebo or Nitro-aspirin placebo plus aspirin in a random order. Primary efficacy variables were changes in urinary albumin excretion (UAE) and in insulin activity at the end of Nitro-aspirin treatment as compared to baseline. UAE (mean of three overnight urine collection), insulin sensitivity (glucose disposal rate as measured by an hyperinsulinemic euglycemic clamp), cardiac haemodynamics (evaluated by echocardiography), NO bioavailability and oxidative stress (measured as nitrite/nitrate plasma levels) and other clinical and laboratory variables, were measured at baseline and at the end of each treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients affected by type 2 diabetes with stable metabolic control (HbA1c < 9%), and stable systemic blood pressure control (SBP/ DBP < 160/90 mmHg).
* Presence of early nephropathy (overnight albumin excretion rate > 20 microg/ min for at least 6 months), without overt renal insufficiency (serum creatinine concentration < 2 mg/dl).
* Age between 18 and 75 years.
* Written signed informed consent; patient willing and able to comply with all study procedures and scheduled visits.

Exclusion Criteria:

* History of any form of allergic reactions or hypersensitivity or intolerance or contraindication to acetylsalicylic acid or nitrates.
* Patients under the age of 18 or above 75.
* Patients who are not able to give an informed consent or inadequate comprehension of study risks and requirements.
* Patients who are unable to comply with the requirements of the study protocol.
* Chronic alcohol or drug abuse (current or within the past year).
* Pregnancy and lactation.
* If women of child-bearing potential, a pregnancy test must be performed before inclusion and after the study, and reliable contraceptive methods followed.
* Evidence for non-diabetic renal disease.
* Patients with duodenal/gastric ulcer history, or gastrointestinal bleeding over the last 6 months.
* Patients with liver insufficiency (ASAT, ALAT > 2 times the upper normal limit).
* Patients with platelet counts < 100,000 cells/mm3.
* Patients with hemorrhagic diathesis.
* Patients on antiinflammatory or immunosuppressive therapy over the last 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13
Dates: Start 2003-03; Study Completion 2004-08

PRIMARY OUTCOMES:
Albuminuria after 4 weeks of treatment
Insulin sensitivity after 4 weeks of treatment
Cardiac and renal hemodynamics after 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Piero Ruggenenti, MD, Principal Investigator — Mario Negri Institute
Locations (1):
- Clinical Research Center for Rare Diseases, Ranica, Bergamo, Italy